CLINICAL TRIAL: NCT03638700
Title: Comparison of the Use of Two High Performance Guidewires in Patients With Stenosis of the Bile Ducts in ERCP: A Randomised Multicenter Trial
Brief Title: Comparison of Two High Performance Guidewires in ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: Klinikum Stadt Hanau (Other); Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor (Other); Robert Bosch Medical Center (Other)
Responsible Party: Principal Investigator, Jorg Albert, Prof. Dr., Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 39/16
Record Dates: First submitted 2016-06-13; First posted 2018-08-20 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Stenosis of Bile Duct
Keywords: stenosis; bile duct; guidewire; ercp
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- guidewire type 1: VisiGlide™ angled tip (Active Comparator): Primary use of VisiGlide™ guidewire (angled tip). In case it should not be possible to complete one step toward the therapeutic goal after 8 to max. 12 minutes after start of the examination, the wire system is changed: primary change to VisiGlide™ (straight tip) resp. to VisiGlid2e™ (tip according to the examiner)
  Interventions: Device: VisiGlide™ angled tip; Device: VisiGlide2™ angled tip; Device: VisiGlide™ straight tip; Device: VisiGlide2™ straight tip
- guidewire type 2: VisiGlide2™ angled tip (Active Comparator): Primary use of VisiGlide2™ guidewire (straight tip). In case it should not be possible to complete one step toward the therapeutic goal after 8 to max. 12 minutes after start of the examination, the wire system is changed: primary change to VisiGlide2™ (angled tip) resp. to VisiGlide™ (tip according to the examiner)
  Interventions: Device: VisiGlide™ angled tip; Device: VisiGlide2™ angled tip; Device: VisiGlide™ straight tip; Device: VisiGlide2™ straight tip
- guidewire type 1: VisiGlide™ straight tip (Active Comparator): Primary use of VisiGlide™ guidewire (straight tip). In case it should not be possible to complete one step toward the therapeutic goal after 8 to max. 12 minutes after start of the examination, the wire system is changed: primary change to VisiGlide™ (angled tip) resp. to VisiGlide2™ (tip according to the examiner)
  Interventions: Device: VisiGlide™ angled tip; Device: VisiGlide2™ angled tip; Device: VisiGlide™ straight tip; Device: VisiGlide2™ straight tip
- guidewire type 2: VisiGlide2™ straight tip (Active Comparator): Primary use of VisiGlide2™ guidewire (straight tip). In case it should not be possible to complete one step toward the therapeutic goal after 8 to max. 12 minutes after start of the examination, the wire system is changed: primary change to VisiGlide2™ (angled tip) resp. to VisiGlide™ (tip according to the examiner)
  Interventions: Device: VisiGlide™ angled tip; Device: VisiGlide2™ angled tip; Device: VisiGlide™ straight tip; Device: VisiGlide2™ straight tip

INTERVENTIONS:
Device: VisiGlide™ angled tip — Arm A: Primary use of VisiGlide™ guidewire (angled tip). In case it should not be possible to complete one step toward the therapeutic goal after 8 to max. 12 minutes after start of the examination, the wire system is changed: primary change to VisiGlide™ (straight tip) resp. to VisiGlid2e™ (tip according to the examiner)
Device: VisiGlide2™ angled tip — Arm B: Primary use of VisiGlide2™ guidewire (angled tip). In case it should not be possible to complete one step toward the therapeutic goal after 8 to max. 12 minutes after start of the examination, the wire system is changed: primary change to VisiGlide2™ (straight tip) resp. to VisiGlide™ (tip according to the examiner)
Device: VisiGlide™ straight tip — Arm C: Primary use of VisiGlide™ guidewire (straight tip). In case it should not be possible to complete one step toward the therapeutic goal after 8 to max. 12 minutes after start of the examination, the wire system is changed: primary change to VisiGlide™ (angled tip) resp. to VisiGlide2™ (tip according to the examiner)
Device: VisiGlide2™ straight tip — Arm D: Primary use of VisiGlide2™ guidewire (straight tip). In case it should not be possible to complete one step toward the therapeutic goal after 8 to max. 12 minutes after start of the examination, the wire system is changed: primary change to VisiGlide2™ (angled tip) resp. to VisiGlide1™ (tip according to the examiner)

SUMMARY:
In ERCP guidewires are used for the insertion of endoprostheses and the cannulation of stenosis. This leads to two essential requirements for the wire systems: The use of a (highly) flexible, hydrophilic wire to achieve successful and rapid passage of the narrow passage; for additional intervention, modern wires are equipped with a stable shaft with which e.g. bougies, dilatation catheters, or stents can be introduced. Guidewires are available with angled or straight tips whose use differ regionally. Guidewires with angled tips are used predominantly in Japan, whereas in the Western world incl. Germany straight wires are commonly used. In a recently published study examining the intubation of the native papilla, successful intubation of the papilla was faster with guidewires with angled tips than with guidewires with straight tips. However, this did not result in an effect upon the time-independent rate of the successful papilla intubation.

The investigators test the hypothesis that 1) a higher success rate of the ERCP can be achieved with the use of an angled guidewire than with a straight guidewire and 2) a higher success rate of the ERCP can be achieved with the use of a type 1 guidewire than with a type 2 guidewire

DETAILED DESCRIPTION:
This is a randomized, multicentric study.

ELIGIBILITY:
Inclusion Criteria:

* Obstruction of the biliary tract (cross sectional imaging or ultrasonography/lab data

Exclusion Criteria:

* Operatively alternated anatomy of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2016-05; Primary Completion 2019-10 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Number of successful passages of bilary (pancreatic) stenosis with the different guidewires. | through study completion, an average of 2 years

SECONDARY OUTCOMES:
Duration of ERCP session | through study completion, an average of 2 years
  Comparison of time needed for the ERCP session in all study groups

CONTACTS AND LOCATIONS:
Overall Officials: Jörg G Albert, Principal Investigator — Robert Bosch Krankenhaus Stuttgart, Germany
Locations (1):
- Goethe University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No